CLINICAL TRIAL: NCT06738056
Title: Real-World Evidence (RWE) Data Analysis of 3-year Usage of Nerivio, a Remote Electrical Neurostimulation (REN) Device In Patients With Migraine
Brief Title: Nerivio Long-term Usage in Patients With Migraine
Status: Completed | Type: Observational
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Other Study IDs: RWE-008
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-04

CONDITIONS: Migraine; Acute Treatment of Migraine
Keywords: Nerivio; Remote Electrical Neuromodulation; Long term usage
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Nerivio users: Patients with migraine who were prescribed the REN wearable device for the treatment of their migraine and began treating between December 2019 and September 2021
  Interventions: Device: Nerivio

INTERVENTIONS:
Device: Nerivio — Remote electrical neuromodulation (REN) wearable device for the treatment of migraine. The device delivers electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. The treatment is self-administered and controlled by a smartphone application.

SUMMARY:
This is a post-marketing real-world evidence study investigates long-term treatment with the Remote Electrical Neuromodulation (REN) wearable Nerivio device over 3 consecutive years in patients with migraine.

DETAILED DESCRIPTION:
The REN device (Nerivio by Theranica, Israel) is a neuromodulation device approved by the FDA for acute and/or preventive treatment of migraine in patients 8 years old and above. It is a wearable device applied to the upper arm. It stimulates C and Aδ noxious fibers. The REN device is operated by a designated app that is downloaded to the user's phone prior first use of the Nerivio device.

As part of the sign-up process for the Nerivio app, all patients accept the terms of use which specifies that providing personal information is done on their own free will and that their de-identified data may be used for research purposes. Users are not obligated to provide personal information and could treat without providing any feedback. The app includes a secure, personal migraine diary, which enables patients to record and track their migraine and other headaches. At the beginning of each treatment, and again 2 hours after the start of treatment, patients are prompted to record their symptoms, including pain level (none, mild, moderate, severe), functional disability (none, mild limitation, moderate limitation, severe limitation), and an indication of which medications, if any, were taken within that 2-hour time window.

This post-marketing RWE study investigates the safety and efficacy of the Nerivio treatment by analyzing data of patients who used the Nerivio device for consecutive 3 years: the following outcome will be assessed:

Primary endpoint:

1. Lack of Tachyphylaxis - No clinically meaningful change in treatment intensity between years.

Secondary endpoints:

1. Consistent effectiveness - Stable pain relief, freedom from pain, functional disability relief, return to normal function (no disability), and freedom from associated symptoms at 2 hours post-treatment relative to baseline in at least 50% of the treatments between years.
2. Utilization - Stable average number of monthly Nerivio treatments per year between years.
3. Safety and tolerability- Number and severity of device related adverse events.

Together, these four objectives provide a comprehensive evaluation of the long-term tolerability, safety, and efficacy of the Nerivio device using a real-world dataset.

ELIGIBILITY:
Inclusion Criteria:

1. - Users who began treating with the REN wearable device between December 2019 and September 2021.
2. - Users who treated migraine attacks consecutively for 3 years, with at least 9 months per year
3. - Users with at least one treatment recorded in each of the counted months.

Exclusion Criteria:

None

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with migraine (age > 12) using the Nerivio device for the treatment of their migraine.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Long Term Lack of Tachyphylaxis | 3 Years
  No clinically meaningful change in treatment intensity between the years (defined as change of less than 2.5 of treatment intensity units between consecutive years).

SECONDARY OUTCOMES:
Long Term Consistent Pain Relief at 2 Hours Post-treatment | 3 Years
  Constant proportion of subjects reporting relief from headache pain at 2 hours post-treatment in at least 50% of their treatments between the years.
  Pain relief is defined as an improvement from severe or moderate pain at treatment initiation to mild or no pain.
  Pain level is reported using a 4-point Likert scale (0 - No pain, 1 - Mild pain, 2 - Moderate pain,3- Severe pain)
Long Term Consistent Pain Freedom at 2 Hours Post-treatment | 3 Years
  Constant proportion of subjects reporting freedom from headache pain at 2 hours post-treatment in at least 50% of their treatments between the years.
  Pain freedom is defined as the disappearance of pain from severe, moderate, or mild headaches at treatment initiation to no pain 2 hours later.
Long Term Consistent Functional Disability Relief at 2 Hours Post-treatment | 3 Years
  Constant proportion of subjects reporting functional disability at the beginning of the treatment and reported improvement of at least one level of functional disability at 2 hours post-treatment in at least 50% of their treatments between the years.
  Functional disability level is reported using a 4-point Likert scale (0-No limitation, 1-Some limitation, 2-Moderate limitation, 3-Severe limitation)
Long Term Consistent Functional Disability disappearance at 2 Hours Post-treatment | 3 Years
  Constant proportion of subjects reporting functional disability at the beginning of the treatment and reported no functional disability at 2 hours post-treatment in at least 50% of their treatments between the years.
  Functional disability level is reported using a 4-point Likert scale (0-No limitation, 1-Some limitation, 2-Moderate limitation, 3-Severe limitation).
Long Term Consistent Freedom from Associated Symptoms at 2-Hours Post-treatment | 3 years
  Constant proportion of subjects reporting presence of associated symptoms (photophobia, phonophobia, nausea and/or vomiting) at the beginning of the treatment and reporting freedom from associated symptoms at 2 hours post-treatment in at least 50% of their treatments between the years.
  Associated symptoms are reported as present or absent
Long Term Utilization of Nerivio | 3 Years
  Constant average number of monthly Nerivio treatments per year between the years.
Device Related Adverse Events | 3 Years
  Incidence of device-related adverse events reported by subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Theranica Bio-Elewctronics Inc, Bridgewater, New Jersey, United States